CLINICAL TRIAL: NCT03149861
Title: Detection of Clinically Significant Prostate Cancer With 18F-DCFPyL PET/MR
Acronym: PSMA-DOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CAPCR ID:17-5295
Record Dates: First submitted 2017-05-01; First posted 2017-05-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Neoplasm, Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No focal biopsy needed (Experimental): Patients in which PET/MR have found no focal findings, will undergo a systemic biopsy as per standard of care, without specific cores for study purposes (Systemic TRUS guided biopsy)
  Interventions: Procedure: Systemic TRUS guided biopsy
- Focal biopsy (Experimental): Patients with a suspicious focal finding on PET/MR, will undergo systemic+focal or focal fusion biopsy (PET/MR-ultrasound guided Fusion biopsy)
  Interventions: Procedure: PET/MR-ultrasound guided Fusion biopsy

INTERVENTIONS:
Procedure: PET/MR-ultrasound guided Fusion biopsy — All focal lesion with PI-RADS >=3 on MR or with DCFPyL uptake on PET will undergo a focal fusion biopsy
  Arms: Focal biopsy
Procedure: Systemic TRUS guided biopsy — Transrectal ultrasound guided systemic prostate biopsy
  Arms: No focal biopsy needed

SUMMARY:
Background:

Currently, patients suspected of having prostate cancer undergo ultrasound-guided systematic biopsies of the prostate. However, up to a quarter of clinically significant tumors, which may pose a risk to patient's well-being, may be missed on random biopsies. MRI enables detection of further tumors in this patient population, but also has limited accuracy.

Study hypothesis:

We hypothesize that hybrid PET-MRI, a novel scanner which incorporates MRI with molecular imaging will improve the detection rate of clinically significant tumors.

Study design:

In this prospective trial, we will recruit 57 men who are suspected of having prostate cancer but have had negative systematic biopsies, who have been diagnosed with low-risk disease but have clinically signs of more aggressive tumor or who have a focal tumor detected and are candidates for minimally-invasive tumor ablation (=tumor destruction with laser or ultrasound waves), in whom it is crucial to exclude other tumor sites.

All patients will undergo PET/MRI after injection of a radiopharmaceutical called "18F-DCFPyL". This is a radioactive probe which has been shown in preliminary studies to be sensitive and specific for detection of prostate cancer.

All lesions detected on PET/MRI will undergo biopsy under ultrasound using fused PET/MRI and ultrasound images for guidance, and compared to histopathology. The primary outcome measure in this study is the proportion of clinically significant prostate cancers that are detected with PET/MRI compared to MRI alone. Improved detection of clinically significant prostate cancer may enable a tailored, personalized therapeutic approach, decreasing morbidity and potentially improving overall patient outcome.

DETAILED DESCRIPTION:
Prostate cancer overview:

Prostate cancer (PCa) is the 3rd leading cause of death from cancer in men and constitutes almost 1/4 of all new cancer cancers in men. Although PCa is prevalent, the risk of clinical or fatal PCa in a 50 year old man is estimated at only 10% and 3%, respectively Currently, over 2/3 of men diagnosed with PCa are diagnosed with organ confined, low risk disease (PSA < 10 ng/ml, Gleason score (=GS) 3+3, cT1c). Management is depending on tumor grade, size and stage and clinical parameters (e.g. life expectancy) and may range from active surveillance to radical therapy including definitive whole gland treatment (radical prostatectomy (RP), or radiotherapy). Although radical whole gland therapy is effective from an oncological standpoint, it may be associated with significant side effects. A more conservative approach in select patients may be enrollment in an active surveillance program. The concept behind this approach is that small volume, low grade PCa may have an indolent course and may not progress to biological significance in the absence of treatment in the patient's lifetime.

Conventional workup of patients with clinical suspicion of PCa:

Transrectal Ultrasound (TRUS)-guided biopsies: Current workup of patients with clinical suspicion of PCa includes TRUS-guided systematic biopsies. These are associated with a relatively high false negative rate, especially for areas difficult to access for biopsy, with csPCa missed in approximately 1 of 4 patients. Furthermore, there is only ˜50% correlation between biopsy obtained GS and final pathology at RP, with upgrading in more than 1 in 3 cases. This may lead to inaccurate risk stratification and inappropriate selection of therapy.

Role of multiparametric-MR & MR-Ultrasound Fusion Biopsy:

In recent years, multiparametric MR (mpMR) has been incorporated in the workup of patients with suspected PCa. T2- weighted imaging (T2WI) in combination with diffusion-weighted imaging (DWI) and dynamic contrast enhanced (DCE)-MR have shown promise in the detection, local staging and risk stratification of PCa, with a reported sensitivity and specificity of 0.74 & 0.88, respectively. Prostate MR is interpreted using a 5-point scoring scale (PI-RADS - Prostate Imaging and Reporting Archiving Data System), with an overall sensitivity & specificity of 77.0% & 71.4%, respectively, for detection of csPCa using PI-RADS-v2. Using MR-US fusion targeted biopsy for mpMR detected lesions improves detection of csPCa compared to standard biopsy (median: 9.1%) and improves correlation of biopsy-derived and surgical tumor grade.

Focal ablation therapy:

In recent years, trials have evaluated various focal ablative therapies (FT) as alternative management for select patients with low/ intermediate risk, organ-confined disease. FT for PCa involves varying degrees of predefined subtotal glandular ablation using a myriad of ablative energy sources e.g high intensity focused ultrasound (HIFU), or laser ablation. The common aim of all of these methods is curative-intent tumor ablation while minimizing morbidity, thereby potentially providing the best balance between oncologic control and side effects of radical therapy. FT relies on the notion that the index lesion can be identified by mpMRI, and localized for intervention. Although no long term data exists on the safety and oncologic outcome of FT, FT appears well-tolerated and associated with significantly less morbidity than whole-gland treatment. At our institution, in-bore focal laser ablation program (MRgFLT) allows patients with a single site of csPCa to be treated while the in-bore HIFU program allows inclusion of patients with up to 2 sites of csPCa confirmed on MR-TRUS fusion biopsy.

One of the main risks with a strategy of FT in PCa is selection failure. Although data is scarce, residual or unrecognized cancer was detected on follow-up biopsy in 22-50% of patients from two separate small series, including cancers in portions of the prostate not appreciated prior to intervention. Although it is uncertain how many of these are csPCa, this highlights the potential limitations of current workup algorithms for patients considered for FT. As only recognized index tumor site is targeted, detection of any further site of csPCa is paramount for appropriate patient selection and therapy success.

Molecular imaging in PCa:

There are shortcomings of current workup of patients with clinical suspicion of PCa, including significant false negative rate of TRUS-biopsies and mpMR. At least 1 in 5 patients in active surveillance program thought to have low-risk disease based on biopsies, turns out to have unfavorable features on surgical pathology. As specific patient management is based on accurate risk stratification, there is a clinical need for further tools to improve identification and characterization of csPCa. There has been increasing interest in molecular imaging in PCa in recent years. The most common radiopharmaceuticals used include choline (11C-Choline/ 18F-Fluorocholine) and 68Ga-PSMA.

PSMA, a type II transmembrane protein, is expressed in normal prostate epithelium and highly expressed in ~90% primary PCa and metastases. 68Ga-PSMA-HBED-CC, the most common PSMA PET radiopharmaceutical assessed to date, has shown high sensitivity in detecting recurrent disease. Recently developed 18F-labelled PSMA compounds (e.g. 18F-DCFPyL) offer several technical advantages over 68Ga including high imaging statistic and higher image resolution. Initial preclinical studies have shown favorable tissue binding and the first clinical investigation in 9 patients has shown very high levels of uptake in primary tumors and metastases with further pilot data suggesting additional metastases identified in >20% of patients compared to 68Ga-PSMA.

Recently introduced hybrid PET/MR scanners allow simultaneous acquisition of MR & PET data, incorporation the advantages of MR and molecular imaging. Emerging data is showing PET/MR to be potentially robust for assessment of oncology indications, particularly those that are better addressed with MR such as PCa. A recently published trial on 68Ga-PSMA PET/MR in intermediate-high risk patients has shown that mpMR, PET and PET/MR had a sensitivity of 66%, 92% and 98%, respectively in localizing Pca. PSMA-PET may also help characterize equivocal lesions on mpMR (PI-RAD v.2 score 3) and may facilitate targeted fusion biopsies of lesions not seen on MR.

ELIGIBILITY:
Inclusion Criteria:

* Patients accrued will fit any of the following criteria:

  1. Clinical suspicion of PCa with negative TRUS-guided biopsy or clinically discordant low-risk PCa (suspicion of more extensive/aggressive disease).
  2. Potential candidates for FT (as per institutional guidelines).

Exclusion Criteria:

Patients will be ineligible to participate in this study if they meet any of the following criteria:

1. Contraindication for MR as per current institutional guidelines.
2. Contraindication for Gadolinium injection as per current institutional guidelines.
3. Inability to lie supine for at least 60 minutes.
4. Prostate biopsy <8 weeks prior to planned PET-MR.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer study
Enrollment: 56 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of clinically significant prostate cancer (csPCa) detected in the study population by 18F-DCFPyL-PET/mpMR as compared to mpMR alone | Through study completion, up to 2 years
  We will compare rates of csPCa detection in 18F-DCFPyL-PET, mpMR and fused 18F-DCFPyL-PET/mpMR, with histopathology obtained at targeted fused US-PET/MR biopsy as the standard of reference

SECONDARY OUTCOMES:
Change in eligibility for focal therapy according to each modality | Through study completion, up to 2 years
  We will document the proportion of patients who meet eligibility criteria for focal therapy, according to each modality (mpMR, 18F-DCFPyL PET and 18F-DCFPyL PET/MR), as determined in consensus between a radiologist and urologist. The change in proportions of eligible patients, according to each modality, will be reported
Correlation of tumor grade to PSMA expression on PET (SUV). | Through study completion, up to 2 years
  Correlation of tumor grade to PSMA expression on PET (SUV).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mirshahvalad SA, Basso Dias A, Ortega C, Abreu Gomez JA, Krishna S, Perlis N, Berlin A, van der Kwast T, Jhaveri K, Ghai S, Metser U, Santiago AT, Veit-Haibach P. [18F]F-DCFPyL PET/MRI radiomics for intraprostatic prostate cancer detection and metastases prediction using whole-gland segmentation. Br J Radiol. 2025 Oct 1;98(1174):1606-1614. doi: 10.1093/bjr/tqaf014. PMID 39847533
- [Derived] Basso Dias A, Ghai S, Ortega C, Mirshahvalad SA, Perlis N, Berlin A, Avery L, Veit-Haibach P, van der Kwast T, Metser U. Impact of 18F-DCFPyL PET/MRI in Selecting Men With Low-/Intermediate-Risk Prostate Cancer for Focal Ablative Therapies. Clin Nucl Med. 2023 Oct 1;48(10):e462-e467. doi: 10.1097/RLU.0000000000004819. PMID 37682613
- [Derived] Metser U, Ortega C, Perlis N, Lechtman E, Berlin A, Anconina R, Eshet Y, Chan R, Veit-Haibach P, van der Kwast TH, Liu A, Ghai S. Detection of clinically significant prostate cancer with 18F-DCFPyL PET/multiparametric MR. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3702-3711. doi: 10.1007/s00259-021-05355-7. Epub 2021 Apr 12. PMID 33846845